CLINICAL TRIAL: NCT02339246
Title: A Steady-state Pharmacokinetic Comparison Of All FK-506 Formulations
Brief Title: Pharmacokinetic Comparison Of All FK-506 Formulations
Acronym: ASTCOFF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Envarsus 3006
Record Dates: First submitted 2014-12-19; First posted 2015-01-15 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-11

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prograf vs Envarsus XR vs Astagraf XL (Active Comparator): Prograft capsules Twice daily for 7 days, followed by Envarsus XR tablets once daily for 7 days followed by Astagraf XL capsules once daily for 7 days.
  Interventions: Drug: Prograf vs Envarsus XR vs Astagraf XL
- Prograf vs Astagraf XL vs Envarsus XR (Active Comparator): Prograf capsules twice daily for 7 days followed by Astagraf XL capsules once daily for 7 days followed by Envarsus XR tablets once daily.
  Interventions: Drug: Prograf vs Astagraf XL vs Envarsus XR

INTERVENTIONS:
Drug: Prograf vs Envarsus XR vs Astagraf XL — prograf vs Envarsus XR vs Astagraf XL
  Other Names: Tacrolimus
  Arms: Prograf vs Envarsus XR vs Astagraf XL
Drug: Prograf vs Astagraf XL vs Envarsus XR — Prograf vs Astagraf XL vs Envarsus XR
  Other Names: Tacrolimus
  Arms: Prograf vs Astagraf XL vs Envarsus XR

SUMMARY:
The purpose of the study is to compare the pharmacokinetic parameters of three different formulations of tacrolimus.

Eligible patients will be treated with all three formulations in a pre-defined sequence.

DETAILED DESCRIPTION:
The pharmacokinetic parameters T(max), C(max) and AUC(0-24) will be compared between the three formulations Envarsus XR once daily, Astagraf XL once daily and Prograf Twice daily.

ELIGIBILITY:
Inclusion Criteria:

1. Renal transplant recipients, males or females, of 18 years of age or above.
2. Able to participate and willing to give written informed consent and to comply with study visits and restrictions.
3. Able to understand English.
4. Patients having received a primary or secondary renal transplant

Exclusion Criteria:

1. Evidence of acute rejection episode within the past three months prior to screening.
2. Recipients of organ transplants other than kidney.
3. Patients who are known to be HIV positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Alloway, PharmD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Philosophe B, Leca N, West-Thielke PM, Horwedel T, Culkin-Gemmell C, Kistler K, Stevens DR. Evaluation of Flexible Tacrolimus Drug Concentration Monitoring Approach in Patients Receiving Extended-Release Once-Daily Tacrolimus Tablets. J Clin Pharmacol. 2018 Jul;58(7):891-896. doi: 10.1002/jcph.1082. Epub 2018 Feb 20. PMID 29462506
- [Derived] Tremblay S, Nigro V, Weinberg J, Woodle ES, Alloway RR. A Steady-State Head-to-Head Pharmacokinetic Comparison of All FK-506 (Tacrolimus) Formulations (ASTCOFF): An Open-Label, Prospective, Randomized, Two-Arm, Three-Period Crossover Study. Am J Transplant. 2017 Feb;17(2):432-442. doi: 10.1111/ajt.13935. Epub 2016 Aug 2. PMID 27340950

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 32 patients were screened (enrolled) and 31 were randomized to treatment.
Groups:
- Envarsus XR: Envarsus XR tablets once daily.
- Astagraf XL: Astagraf XL capsules once daily.
- Prograf: Prograf capsules twice daily.
Period: First Intervention (7 Days)
Arm/Group | Envarsus XR | Astagraf XL | Prograf
Started | 0 | 0 | 31
Completed | 0 | 0 | 31
Not Completed | 0 | 0 | 0
Period: Second Intervention (7 Days)
Arm/Group | Envarsus XR | Astagraf XL | Prograf
Started | 16 | 15 | 0
Completed | 16 | 15 | 0
Not Completed | 0 | 0 | 0
Period: Third Period (7 Days)
Arm/Group | Envarsus XR | Astagraf XL | Prograf
Started | 15 | 16 | 0
Completed | 15 | 16 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prograf vs Envarsus XR vs Astagraf XL: Prograft capsules Twice daily Envarsus XR tablets once daily Astagraf XL capsules once daily
  Prograf vs Envarsus XR vs Astagraf XL: prograf vs Envarsus XR vs Astagraf XL
- Prograf vs Astagraf XL vs Envarsus XR: Prograf capsules twice daily Astagraf XL capsules once daily Envarsus XR tablets once daily
  Prograf vs Astagraf XL vs Envarsus XR: Prograf vs Astagraf XL vs Envarsus XR
- Total: Total of all reporting groups
Arm/Group | Prograf vs Envarsus XR vs Astagraf XL | Prograf vs Astagraf XL vs Envarsus XR | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (11.00) | 46.3 (13.30) | 48.3 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of T(Max) for Envarsus XR, Astagraf XL and Prograf.
Description: Tacrolimus whole blood concentrations obtained from the central lab was used for PK analysis. Actual sampling times was used to calculate T(max).
  Nominal time points used were:
  Prograf sampling strategy (21 samples): Pre-dose (C0) and then 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 12.5, 13, 13.5, 14, 14.5, 15, 16, 18, 20, and 24.
  Envarsus XR sampling strategy (18 samples): Pre-dose (C0) and then 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 18, 21, 24, and 27.
  Astagraf XL sampling strategy (17 samples): Pre-dose (C0) and then 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 18, 21, and 24.
Time Frame: 8 days
Population: One patient in the Envarsus XR arm was excluded from the analysis due to non compliance.
Measure: Median (95% Confidence Interval); unit: hour
Arm/Group | Envarsus XR | Astagraf XL | Prograf
Number analyzed (Participants) | 30 | 30 | 30
hour | 5.91 [1.45 to 13.95] | 1.93 [0.92 to 5.92] | 1.48 [0.93 to 19.97]

2. Primary Outcome: Evaluation of C(Max) for Envarsus XR, Astagraf XL and Prograf.
Description: Tacrolimus whole blood concentrations obtained from the central lab was used for PK analysis. Actual sampling times was used to calculate C(max).
  Nominal time points used were:
  Prograf sampling strategy (21 samples): Pre-dose (C0) and then 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 12.5, 13, 13.5, 14, 14.5, 15, 16, 18, 20, and 24.
  Envarsus XR sampling strategy (18 samples): Pre-dose (C0) and then 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 18, 21, 24, and 27.
  Astagraf XL sampling strategy (17 samples): Pre-dose (C0) and then 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 18, 21, and 24.
Time Frame: 8 days
Population: One patient in the Envarsus XR arm was excluded from the analysis due to non compliance.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Envarsus XR | Astagraf XL | Prograf
Number analyzed (Participants) | 30 | 30 | 30
ng/mL | 13.88 (5.331) | 13.17 (12.49) | 14.54 (13.60)

3. Primary Outcome: Evaluation of AUC(0-24) for Envarsus XR, Astagraf XL and Prograf.
Description: Tacrolimus whole blood concentrations obtained from the central lab was used for PK analysis. Actual sampling times was used to calculate AUC(0-24).
  Nominal time points used were:
  Prograf sampling strategy (21 samples): Pre-dose (C0) and then 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 12.5, 13, 13.5, 14, 14.5, 15, 16, 18, 20, and 24.
  Envarsus XR sampling strategy (18 samples): Pre-dose (C0) and then 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 18, 21, 24, and 27.
  Astagraf XL sampling strategy (17 samples): Pre-dose (C0) and then 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 18, 21, and 24.
Time Frame: 8 days
Population: One patient in the Envarsus XR arm was excluded from the analysis due to non compliance.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Envarsus XR | Astagraf XL | Prograf
Number analyzed (Participants) | 30 | 30 | 30
hr*ng/mL | 213.41 (83.095) | 165.02 (48.910) | 176.52 (50.799)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of first dose of study drug and until last visit which was approximately 1 month.
Groups:
- Astagraf XR: Astagraf XR capsules once daily.
Arm/Group | Envarsus XR | Astagraf XR | Prograf
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 2/31 | 10/31 | 3/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Envarsus XR (N=31) | Astagraf XR (N=31) | Prograf (N=31)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days